CLINICAL TRIAL: NCT00000909
Title: A Randomized, Open Label Phase II Study of Subcutaneous Interleukin-2 (Proleukin) Alone vs No Therapy in Patients With HIV Infection and at Least 350 CD4+ Cells/mm3 Who Do Not Wish to Receive Treatment With Antiretroviral Therapy
Brief Title: A Study to Evaluate the Effects of Giving IL-2 Alone to HIV-Positive Patients With CD4 Cell Counts of at Least 350 Cells/mm3 Who Do Not Wish to Receive Anti-HIV Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRP 021D; 10462 (Registry Identifier: DAIDS ES); IL-2 UK
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Interleukin-2; Dose-Response Relationship, Drug; CD4 Lymphocyte Count; RNA, Viral
MeSH Terms: conditions — HIV Infections | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of giving interleukin-2 (IL-2) alone to HIV-positive patients with CD4 cell counts greater than 350 cells/mm3 who do not wish to receive anti-HIV (antiretroviral) therapy. This study will also determine if IL-2 given alone can increase CD4 cell counts or decrease the level of HIV in the blood.

IL-2 (a protein found in the blood that helps boost the immune system) can result in increases in CD4 cell count (immune system cells that fight infection). IL-2 is normally given in combination with antiretroviral therapy to treat HIV infection; however, some HIV patients do not wish to take antiretrovirals. This study asks if it is safe and effective to take IL-2 alone to treat HIV infection.

DETAILED DESCRIPTION:
Previous studies have shown that interleukin-2, when given under the skin, results in CD4+ cell count increases, and may impact upon disease progression. A Phase III trial is the next step in the development of these efficacy trials. One question, however, has not been addressed in previous IL-2 studies: whether it is both safe and reasonable to allow prospective IL-2 recipients the autonomy of choosing whether or not to take antiretrovirals in addition to their cytokine therapy. This trial addresses that concern.

In this open-label study, 36 patients are randomized to 1 of 3 treatment groups of 12 patients each:

Group I: IL-2 every 12 hours for 5 days every 8 weeks. Group II: IL-2 every 12 hours for 5 days every 8 weeks (higher IL-2 dose). Group III: Control group receiving no therapy. Patients must complete a minimum of 3 8-week cycles of treatment. Twelve patients are randomized to each arm. Following study completion, Group I and II patients may elect to continue receiving IL-2 during follow-up or as part of an additional protocol based on the results of this study.

[AS PER AMENDMENT 2/12/99: Patients who have received study medication and/or routine protocol visits and procedures for at least 6 months with acceptable compliance are eligible for continued follow-up in an extension phase. The extension phase will continue for at least 1 year from the date when the last patient has been enrolled in the extension phase. Patients originally randomized to IL-2 may continue to receive IL-2 during the extension period, with IL-2 therapy guided on an individual basis. Patients originally randomized to no therapy may continue to receive no therapy during the extension phase.] [AS PER AMENDMENT 7/11/00: Patients demonstrating acceptable compliance with routine visits and procedures during the initial treatment phase and/or extension phase may participate in the long-term follow-up phase which requires follow-up visits at least every 4 months for approximately 5 years. Patients originally randomized to Group 1 or 2 may continue to receive IL-2, with IL-2 therapy guided on an individual basis, during the long-term follow-up phase. Patients originally randomized to Group 3 may continue to receive no therapy during the long-term follow-up phase.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have had at least one CD4 cell count greater than or equal to 350 cells/mm3 within 30 days of study entry.
* Are at least 18 years old.
* Agree to abstinence or use of effective methods of birth control 1 month before and during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a history of a potentially life-threatening autoimmune or inflammatory disease.
* Abuse alcohol or drugs, or have any serious psychiatric or medical illnesses that would affect their safety or ability to complete the study.
* Have a history of an AIDS-defining illness.
* Have a history of cancer, other than Kaposi's sarcoma.
* Have ever taken IL-2 or any antiretroviral medications.
* Are pregnant.
* Are taking certain medications, including anti-seizure medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Youle, Study Chair; Jorge Tavel, Study Chair
Locations (1):
- Kobler Ctr. of Chelsea Westminster Hosp. C604-030 CRS, London, United Kingdom